CLINICAL TRIAL: NCT02765841
Title: A Phase 3, Single-arm, Open-label, International, Multi-center Study to Evaluate the Efficacy and Safety of Lomitapide in Pediatric Patients With Homozygous Familial Hypercholesterolemia on Stable Lipid-lowering Therapy
Brief Title: Evaluate the Efficacy and Safety of Lomitapide in Pediatric Patients With Homozygous Familial Hypercholesterolemia on Stable Lipid-lowering Therapy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEGR-733-020
Record Dates: First submitted 2016-04-27; First posted 2016-05-09 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Homozygous Familial Hypercholesterolemia
Keywords: HoFH
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — BMS201038

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lomitapide (Experimental)
  Interventions: Drug: Lomitapide

INTERVENTIONS:
Drug: Lomitapide
  Other Names: Juxtapid, Lojuxta

SUMMARY:
This is a Phase 3 single-arm, open-label, international, multi-center clinical trial to evaluate the efficacy and safety of lomitapide in pediatric patients with HoFH who are receiving stable lipid-lowering therapy, including LDL apheresis. The study is comprised of a 12-week Run-in Period, a primary 24-week Efficacy Phase, followed by an 80-week Safety Phase.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥5 and <18 years with diagnosed functional HoFH
2. Patient must weigh at least 15 kg and be at or above the 10th percentile in BMI and at least 10th percentile in height for age and gender based on CDC growth charts
3. Negative pregnancy test at Screening and during the study for females of child bearing age
4. Potentially sexually active female patients who are of child-bearing age must either be sexually abstinent or follow two acceptable methods of contraception

Exclusion Criteria:

1. Other forms of primary hyperlipoproteinemia and secondary causes of hypercholesterolemia (e.g., nephrotic syndrome, hypothyroidism).
2. Abnormal liver function test at Screening
3. Moderate or severe hepatic impairment or active liver disease
4. Serum creatine phosphokinase (CPK) level >2 × ULN.
5. Chronic renal insufficiency
6. History of drug abuse within the last 3 years or habitual alcohol consumption
7. New York Heart Association (NYHA) Class III or IV congestive heart failure.
8. Uncontrolled hypertension
9. In the judgment of the PI, precocious or delayed puberty or endocrine disorder that would affect growth
10. History of non-skin malignancy or other cancers occurring within the past 3 years
11. History of inflammatory bowel disease or other malabsorption syndrome or a history of bowel resection, gastric bypass, or other weight loss surgical procedure.
12. Use of mipomersen within 6 months of Screening.
13. Any medical condition for which the life expectancy is predicted to be less than 5 years.
14. Any patient who is unable to avoid treatment with strong or moderate cytochrome P450 3A4 (CYP3A4) inhibitors, or other drugs contraindicated for use with lomitapide during the study.
15. Participation in an interventional clinical study within 6 weeks for a statin therapy or within 6 months for any other unapproved therapy.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Percent change in LDL-C | Baseline, Week 24

SECONDARY OUTCOMES:
Percent Change in TC | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 68, 80, 92, 104
Percent change in non-HDL-C | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 68, 80, 92, 104
Percent change in HDL-C | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 68, 80, 92, 104
Percent change in TG | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 68, 80, 92, 104
Percent change in VLDL-C | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 68, 80, 92, 104
Percent change in Lp(a) | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 68, 80, 92, 104
Percent change in apo B | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 68, 80, 92, 104
Percent change in apo A-1 | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 68, 80, 92, 104
Percent change in LDL-C | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 68, 80, 92, 104
Changes in lipid-lowering therapy | Week 24 through Week 104
Changes in LDL apheresis | Week 24 through Week 104
Percent of patients achieving goal (LDL-C of <100 mg/dL [2.6 mmol/L] for patients without documented cardiovascular disease [CVD] at Baseline | Week 24 and through Week 108
Percent of patients achieving goal LDL-C of <70 mg/dL [1.8 mmol/L]) for patients with documented CVD at Baseline. | Week 24 and through Week 108
Changes in laboratory parameters (including hepatic and renal function) | Baseline through Year 2
Reported Adverse Events | Baseline through Year 2
Electrocardiogram (ECG) changes | Baseline through Year 2
Pulmonary function tests (PFTs) | Baseline through Year 2
Bone health/age (x-ray of the wrist) | Baseline through Year 2
Height Measurement | Baseline through Year 2
Weight Measurement | Baseline through Year 2
Body Mass Measurement | Baseline through Year 2
Tanner Staging | Baseline through Year 2
Percent change in hepatic fat | Baseline through Year 2
Blood Pressure | Baseline through Year 2
Heart Rate | Baseline through Year 2
Temperature | Baseline through Year 2
Respiration (breaths/min) | Baseline through Year 2